CLINICAL TRIAL: NCT00921765
Title: Naloxone Block of Low-dose (Analgetic Dose) Ketamine
Brief Title: Reversal of Ketamine Pharmacodynamic Effects With Naloxone
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Problems with patient recruitment
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Lasse Ansgar Skoglund, Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DOK-018
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Pain
Keywords: Pain; Naloxone; Ketamine; Third Molar; Surgery
MeSH Terms: conditions — Pain | interventions — Sodium Chloride; Ketamine; Naloxone

STUDY DESIGN:
Intervention Model Description: Parallell Group design should be used when final dose had been found
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind (one making drug solutions) another administrating the drugs
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo + Placebo (Placebo Comparator): Saline single bolus dose iv + saline single bolus dose iv
  Interventions: Drug: Saline
- Placebo + Ketamine (Active Comparator): Saline single bolus dose followed by single bolus dose of ketamine 0.2 mg/kg bw
  Interventions: Drug: Saline + Ketamine
- Naloxone + Placebo (Active Comparator): Single bolus dose of naloxone 0.2 mg/kg bw followed by single bolus dose of saline
  Interventions: Drug: Naloxone + Placebo
- Naloxone + Ketamine (Active Comparator): Single bolus dose of ketamine 0.2 mg/kg bw followed by single bolus dose of ketamine 0.2 mg/kg bw
  Interventions: Drug: Naloxone + Ketamine

INTERVENTIONS:
Drug: Saline — Saline single bolus dose followed by saline single bolus dose iv
  Other Names: Physiological saline 0.9%
  Arms: Placebo + Placebo
Drug: Saline + Ketamine — Single bolus dose of saline followed by ketamine 0.2 mg/kg bw
  Other Names: Physiological saline 0.9%; Ketamine; ATC code: N01A X03
  Arms: Placebo + Ketamine
Drug: Naloxone + Placebo — Single bolus dose of naloxone 0.2 mg/kg bw followed by single bolus dose of saline
  Other Names: Naloxone; ATC code: V03A B15; Physiological saline 0.9%
  Arms: Naloxone + Placebo
Drug: Naloxone + Ketamine — Single bolus dose of naloxone 0.2 mg/kg bw followed by single bolus dose of ketamine 0.2 mg/kg bw
  Other Names: Naloxone; ATC code: V03A B15; Ketamine; ATC code: N01A X03
  Arms: Naloxone + Ketamine

SUMMARY:
The purpose of this study is to determine whether the analgetic and other effects effect of ketamine are partly mediated through opioid receptors

DETAILED DESCRIPTION:
Ketamine er et dissociative anaesthetic closely related with phencyclidine (PCP). Phencyclidine is a non-competitive NMDA-antagonist, and it is assumed that the pharmacodynamic mechanism of action for ketamine is the same. Receptor binding studies shows that ketamine has affinity to many receptor types, including opioid mu and kappa receptors. Ketamine has only about 25 times lower affinity for kappa receptors than for the NMDA-receptor complex. Naloxone is a specific antagonist for opioid receptors and block both mu og kappa receptors. A dose of naloxone 10 times larger than required to block mu receptors is required to block kappa receptors. Experiments with naloxone suggest that ketamine is not a mu agonist, but experiments with sufficient large naloxone doses to block kappa receptors have not been carried out in humans.

ELIGIBILITY:
Inclusion Criteria:

* Females of norwegian Caucasian origin who needs surgical removal of impacted third molars

Exclusion Criteria:

* Anamnestic information regarding psychiatric diagnosis regarding mother/father or brother/sister Concommitant medication other than oral contraceptives Hypersensitivity towards NSAID/opioids/study drugs Females with suspected or confirmed pregnancy Lactating females Surgery lasting more than 60 minutes

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2009-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity (0-10 Numerical Rating Scale) | 30 minutes

SECONDARY OUTCOMES:
Subjective measurement of psychotomimetic effects | 30 minutes
Adverse effects | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Olav Hustveit, MD, PhD, Study Director — University of Oslo; Elena Landari, DDS, Principal Investigator — University of Oslo
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gear RW, Miaskowski C, Gordon NC, Paul SM, Heller PH, Levine JD. Kappa-opioids produce significantly greater analgesia in women than in men. Nat Med. 1996 Nov;2(11):1248-50. doi: 10.1038/nm1196-1248. PMID 8898754
- [Background] Hustveit O, Maurset A, Oye I. Interaction of the chiral forms of ketamine with opioid, phencyclidine, sigma and muscarinic receptors. Pharmacol Toxicol. 1995 Dec;77(6):355-9. doi: 10.1111/j.1600-0773.1995.tb01041.x. PMID 8835358
- [Background] Mathisen LC, Skjelbred P, Skoglund LA, Oye I. Effect of ketamine, an NMDA receptor inhibitor, in acute and chronic orofacial pain. Pain. 1995 May;61(2):215-220. doi: 10.1016/0304-3959(94)00170-J. PMID 7659431
- [Background] Oye I, Paulsen O, Maurset A. Effects of ketamine on sensory perception: evidence for a role of N-methyl-D-aspartate receptors. J Pharmacol Exp Ther. 1992 Mar;260(3):1209-13. PMID 1312163